CLINICAL TRIAL: NCT00833911
Title: An Open-Label Long-term Safety Study of Tramadol HCl OAD (Once A Day) 300 mg in the Treatment of Pain Due to Osteoarthritis of the Knee
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Labopharm Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDT3-004; NCT00833911 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2009-01-29; First posted 2009-02-02 (Estimated); Results first posted 2009-06-02 (Estimated); Last update posted 2012-04-30 (Estimated); Status verified 2012-04

CONDITIONS: Osteoarthritis, Knee
Keywords: Moderate to severe symptomatic osteoarthritis of the knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tramadol Contramid® OAD (Experimental)
  Interventions: Drug: Tramadol Once A Day

INTERVENTIONS:
Drug: Tramadol Once A Day

SUMMARY:
The purpose of this study is to collect information regarding the long-term (6 and 12 months) safety of Tramadol HCl Once-A-Day(OAD) 300 mg.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female patients between the ages of 40-75 with a diagnosis of Osteoarthritis of the knee consistent with the American College of Rheumatology (ACR) Clinical Classification Criteria for Arthritis of the Knee (Altman, R. et al., 1991):

   * Current knee pain,
   * Less than 30 minutes of morning stiffness with or without crepitus on active motion,
   * Confirmation either by arthroscopy or radiologist's report (X-rays showing osteophytes, joint space narrowing or subchondral bone sclerosis {eburnation}) within two years prior to entry into the study.
2. Erythrocyte Sedimentation Rate (ESR) < 40 mm/hour.
3. Western Ontario and McMaster Osteoarthritis Index (WOMAC) Pain Subscale total score of >= 150 mm at baseline. (5 questions/100 mm scale each with an averaged response of 30 mm or higher per question).
4. Oral and written language comprehension at a level sufficient to comply with the protocol and complete study-related materials.
5. The Patient has signed and dated the Research Ethics Board (REB) approved, written, informed consent prior to study participation.

Exclusion Criteria:

1. Known rheumatoid arthritis or any other rheumatoid disease.
2. Secondary arthritis i.e. any of the following: septic arthritis; inflammatory joint disease; gout; pseudogout; Paget's disease; joint fracture; acromegaly; fibromyalgia; Wilson's disease; Ochronosis; Haemochromatosis; Osteochondromatosis; heritable arthritic disorders; or collagen gene mutations.
3. Obesity Class II (Body Mass Index (BMI) >= 35) (National Institutes of Health (NIH), 2000).
4. Major illness requiring hospitalization during the 3 months before commencement of the screening period.
5. Patients who are unwilling to stop taking pain medication other than the study medication (for arthritis or other types of pain) or are unwilling to stop taking other medications for the treatment of osteoarthritis (OA).
6. Patients who have previously failed tramadol hydrochloride (HCl) therapy or those who discontinued tramadol HCl due to adverse events.
7. Patients who are taking or within the last 3 weeks have taken the following medications: monoamine oxidase inhibitors; tricyclic antidepressants and other tricyclic compounds (e.g. cyclobenzaprine, promethazine); neuroleptics; selective serotonin reuptake inhibitors; or other drugs which reduce seizure threshold.
8. Patients who are taking or have taken another investigational agent within the last 30 days.
9. Patients with a history of seizure disorder other than Infantile Febrile Seizures.
10. Patients who are opioid dependent.
11. Patients with bowel disease causing malabsorption.
12. Patients who are pregnant or lactating or patients of child-bearing potential who are unwilling to utilize a medically approved method of contraception during participation in this clinical trial.
13. Patients with significant liver disease, defined as active hepatitis or elevated liver enzymes >3 times the upper boundary of the normal range.
14. Patients with significant renal disease, defined as creatinine clearance <30 mL/min as estimated by the method of Levey et al., 1999.
15. Current substance abuse or dependence, other than nicotine.
16. Allergy or adverse reaction to tramadol or any structurally similar drugs e.g. opiates.
17. Any other condition that, in the opinion of the investigators, would adversely affect the patient's ability to complete the study or its measures.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Actual)
Dates: Start 2003-04; Primary Completion 2004-07 (Actual); Study Completion 2004-07 (Actual)

REFERENCES:
- [Result] Mongin G. Tramadol extended-release formulations in the management of pain due to osteoarthritis. Expert Rev Neurother. 2007 Dec;7(12):1775-84. doi: 10.1586/14737175.7.12.1775. PMID 18052769
- See also: Approved labelling — http://dailymed.nlm.nih.gov/dailymed/drugInfo.cfm?id=9048

RESULTS

PARTICIPANT FLOW:
Period: Titration
Arm/Group | 300 mg Tramadol HCl OAD
Started | 392
Completed | 371
Not Completed | 21
Not completed — Adverse Event | 18
Not completed — Withdrawal by Subject | 3
Period: Maintenance Phase I
Arm/Group | 300 mg Tramadol HCl OAD
Started | 371
Completed | 273
Not Completed | 98
Not completed — Adverse Event | 73
Not completed — Withdrawal by Subject | 11
Not completed — Physician Decision | 10
Not completed — Lack of Efficacy | 4
Period: Maintenance Phase II
Arm/Group | 300 mg Tramadol HCl OAD
Started | 176 (97 patients chose not to continue into Maintenance Phase II)
Completed | 166
Not Completed | 10
Not completed — Adverse Event | 6
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 1
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Arm/Group | 300 mg Tramadol HCl OAD
Number analyzed (Participants) | 392
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 229
  >=65 years | 163
Age Continuous [Mean (Standard Deviation); unit: years] | 61.4 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 333
  Male | 59

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Having Experienced an Adverse Event During the 6-12 Month Open-Label Safety Participation
Description: Spontaneous reports of adverse events were recorded for the entire study population, the 6-months safety population and the 12-months safety population
Time Frame: 6 months and 12 months
Population: All patients having taken 1 dose of 300 mg Tramadol HCl OAD at a minimum are being assessed for adverse event occurence for up to 12 months.
  6-months safety: patients who completed at least 175 days on treatment.
  12-months safety: patients who completed at least 350 days on treatment.
Measure: Number; unit: participants
Groups:
- All Patients With 1 Dose of 300 mg Tramadol HCl OAD Minimum: All patients in the study who took at least one dose of 300 mg Tramadol HCl OAD. Overall time frame for this population is 0-12 months.
Arm/Group | All Patients With 1 Dose of 300 mg Tramadol HCl OAD Minimum | 6-months Safety | 12-months Safety
Number analyzed (Participants) | 392 | 275 | 168
participants | 346 | 188 | 121

ADVERSE EVENTS:
Arm/Group | All Patients With 1 Dose of 300 mg Tramadol HCl OAD Minimum | 6-months Safety | 12-months Safety
Serious Adverse Events (participants affected / at risk) | 9/392 | 1/275 | 0/168
Other Adverse Events (participants affected / at risk) | 321/392 | 169/275 | 101/168
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients With 1 Dose of 300 mg Tramadol HCl OAD Minimum (N=392) | 6-months Safety (N=275) | 12-months Safety (N=168)
Acute pulmonary oedema (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Cerebrovascular accident (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis, Not Otherwise Specified (NOS) (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetes mellitus, Not Otherwise Specified (NOS) (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis aggravated (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis chronic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Paresis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients With 1 Dose of 300 mg Tramadol HCl OAD Minimum (N=392) | 6-months Safety (N=275) | 12-months Safety (N=168)
Anorexia (Metabolism and nutrition disorders) | 21 (22) | 15 (16) | 8 (8)
Constipation (Gastrointestinal disorders) | 121 (155) | 74 (86) | 40 (51)
Dizziness (Nervous system disorders) | 106 (134) | 30 (42) | 22 (36)
Fatigue (General disorders) | 19 (27) | 15 (20) | 4 (4)
Headache (Nervous system disorders) | 62 (80) | 25 (31) | 28 (42)
Hypertension (Vascular disorders) | 15 (15) | 5 (5) | 10 (10)
Influenza (Infections and infestations) | 19 (22) | 18 (20) | 7 (8)
Nasopharyngitis (Infections and infestations) | 22 (25) | 16 (17) | 13 (15)
Nausea (Gastrointestinal disorders) | 159 (233) | 62 (92) | 42 (67)
Pruritus (Skin and subcutaneous tissue disorders) | 21 (23) | 4 (4) | 1 (1)
Somnolence (Nervous system disorders) | 99 (116) | 29 (36) | 13 (13)
Sweating increased (Skin and subcutaneous tissue disorders) | 23 (25) | 18 (20) | 2 (3)
Urinary tract infection (Infections and infestations) | 20 (20) | 7 (7) | 10 (10)
Vertigo (Ear and labyrinth disorders) | 31 (38) | 8 (9) | 8 (11)
Vomiting (Gastrointestinal disorders) | 55 (67) | 17 (24) | 13 (17)
Weight decreased (Investigations) | 29 (29) | 16 (16) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to submitting results communications, the investigator shall allow Labopharm at least 30 days to review the proposed communication. If the proposed publication/disclosure risks Labopharm's ability to patent any invention related to the study, the publication or disclosure will be modified or delayed to allow Labopharm to seek patent protection. This statement does not give Labopharm any editorial rights other than to restrict the disclosure of Labopharm's confidential information.